CLINICAL TRIAL: NCT02777268
Title: A Single Centre, Open Label, Randomised, Crossover Study in Dexamethasone-suppressed Healthy Adult Male Volunteers to Compare the Pharmacokinetics of Infacort® Versus Immediate-release Hydrocortisone Tablets at a Single Dose of 10 mg and to Evaluate the Dose Proportionality of Infacort® at Doses of 0.5 mg, 2 mg, 5 mg and 10 mg
Brief Title: Comparison of Pharmacokinetics of Infacort® Versus Immediate-release Hydrocortisone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Infacort 001
Record Dates: First submitted 2016-04-27; First posted 2016-05-19 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Infacort 0.5 mg (Experimental): Multi-particulate granules from 1 (0.5 mg) capsule
  Interventions: Drug: Infacort
- Infacort 2 mg (Experimental): Multi-particulate granules from 1 (2 mg) capsule
  Interventions: Drug: Infacort
- Infacort 5 mg (Experimental): Multi-particulate granules from 1 (5 mg) capsule
  Interventions: Drug: Infacort
- Infacort 10 mg (Experimental): Multi-particulate granules from 1 (10 mg) capsule
  Interventions: Drug: Infacort
- Hydrocortisone (Active Comparator): 1 (10 mg) tablet
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Infacort — Multi-particulate granules
  Arms: Infacort 0.5 mg; Infacort 10 mg; Infacort 2 mg; Infacort 5 mg
Drug: Hydrocortisone — Tablet
  Arms: Hydrocortisone

SUMMARY:
This was a single centre, open-label, randomised, 5-way crossover study.

DETAILED DESCRIPTION:
This was a single centre, open-label, randomised, 5-way crossover study design to compare the PK of Infacort® versus immediate-release hydrocortisone tablets and to evaluate the dose proportionality of 0.5 mg, 2 mg, 5 mg and 10 mg Infacort®. The study was conducted in 1 cohort of 16 healthy male subjects and comprised a Screening Visit, 5 treatment periods (Treatment Periods 1 to 5) and a Post-study Visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between 18 and 60 years of age, inclusive (at Screening Visit).
* Subjects with a Body Mass Index (BMI) of 21-28.
* Subjects with no clinically significant abnormal serum biochemistry, haematology and urine examination values within 14 days prior to the first dose of investigational medicinal product (IMP).
* Subjects with a negative urinary drugs of abuse screen determined within 14 days prior to the first dose of IMP. A positive alcohol test may have been repeated at the discretion of the Investigator.
* Subjects with negative human immunodeficiency virus (HIV) and hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results.
* Subjects with no clinically significant abnormalities in 12-lead electrocardiogram (ECG) determined within 14 days prior to the first dose of IMP.
* Subjects with no clinically-significant deviation outside the normal ranges for blood pressure and pulse measurements.
* Subjects (unless anatomically sterile or where abstaining from sexual intercourse was in-line with the preferred and usual lifestyle of the subject) and sexual partners used effective contraception methods during the trial and for 3 months after the last dose of IMP, for example; oral contraceptive + condom, intra-uterine device (IUD) + condom or diaphragm with spermicide + condom.
* Subjects were available to complete the study.
* Subjects satisfied a medical examiner about their fitness to participate in the study.
* Subjects provided written informed consent to participate in the study.

Exclusion Criteria:

* A clinically significant history of gastrointestinal disorder likely to influence drug absorption.
* Receipt of regular medication within 14 days prior to the first dose of IMP (including high dose vitamins, dietary supplements or herbal remedies).
* Receipt of any vaccination within 14 days prior to the first dose of IMP.
* Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
* Presence of clinically significant infections (systemic fungal and viral infections, acute bacterial infections).
* Current or previous history of tuberculosis.
* A clinically significant history of previous allergy / sensitivity to hydrocortisone and/or dexamethasone.
* A clinically significant history or family history of psychiatric disorders/illnesses.
* A clinically significant history of drug or alcohol abuse.
* Inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function).
* Participated in a New Chemical Entity clinical study within the previous 4 months or a marketed drug clinical study within the previous 3 months. (N.B. The washout period between trials was defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
* Subjects who had consumed more than 2 units of alcohol per day within 7 days prior to the first dose of IMP or had consumed any alcohol within the 48 hr period prior to the first dose of IMP.
* Donation of 450 mL or more of blood within the previous 3 months.
* Subjects who smoked (or ex-smokers who had smoked within 6 months prior to first dose of IMP).
* Subjects who worked shifts (i.e. regularly alternated between days, afternoons and nights).

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Girish Sharma, MD, Principal Investigator — Simbec Research

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Area: United Kingdom Location: Phase 1 Unit
Groups:
- All Study Participants: 5-way crossover study design involving Infacort and hydrocortisone at the following dose strengths:
  Infacort 0.5mg Infacort 2mg Infacort 5mg Infacort 10mg Hydrocortisone 10mg
  Each IMP was administered to each subject in a randomised, crossover manner over 5 treatment periods (1 treatment/period). During each treatment period, each subject was admitted to the Unit on the afternoon of Day 1 and remained in the Unit until completion of all scheduled assessments on Day 2. Each subject received their scheduled IMP on the morning of Day 2 at ~0700hrs (fasted). Each subject also received 1mg dexamethasone (to suppress endogenous cortisol production) at approximately 2200hrs on Day 1, and at approximately 0600hrs and 1200hrs on Day 2. All doses were administered with 200mL water. There were at least 7 days washout between each dose of IMP.
Period: Overall Study
Arm/Group | All Study Participants
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.70 (14.370)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — United Kingdom
  participants
    United Kingdom | 16
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.34 (2.085)
Height (m) [Mean (Standard Deviation); unit: Metres (m)] | 1.773 (0.081)
Weight (kg) [Mean (Standard Deviation); unit: Kilograms (kg)] | 79.70 (8.543)
Medical History and Concurrent Conditions [Count of Participants; unit: Participants] | 0
Drug/Alcohol and HIV/Hepatitis Screening [Count of Participants; unit: Participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Infacort vs Hydrocortisone
Description: To compare the Cmax of Infacort® versus immediate-release hydrocortisone in a single dose of 10 mg.
Time Frame: -1h, -0.5h, 0h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 4.5h, 5h, 5.5h, 6h, 6.5h, 7h, 7.5h, 8h, 9h, 10h, 11h, 12h
Population: Two subjects were excluded from the Infacort 10mg analysis population due to inadequate endogenous cortisol suppression prior to dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- Infacort 10mg: Multi-particulate granules from 10mg Infacort capsule
Arm/Group | Infacort 10mg | Hydrocortisone
Number analyzed (Participants) | 14 | 14
nmol/L | 601.843 (21.5) | 622.384 (15.8)

2. Primary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of Infacort vs Hydrocortisone
Description: To compare the Tmax of Infacort® versus immediate-release hydrocortisone in a single dose of 10 mg.
Time Frame: -1h, -0.5h, 0h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 4.5h, 5h, 5.5h, 6h, 6.5h, 7h, 7.5h, 8h, 9h, 10h, 11h, 12h
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: Hour
Groups:
- Infacort 10mg: Multi-particulate granules from a 10mg Infacort capsule.
- Hydrocortisone: 10 mg hydrocortisone tablet
Arm/Group | Infacort 10mg | Hydrocortisone
Number analyzed (Participants) | 14 | 14
Hour | 0.500 (0.4031) | 1 (0.4171)

3. Primary Outcome: Area Under the Curve (AUC0-t) of Infacort vs Hydrocortisone
Description: To compare the AUC0-t of Infacort® versus immediate-release hydrocortisone in a single dose of 10 mg. AUC0-t represents the total exposure to drug over time, hence the reporting of a single value below.
Time Frame: -1h, -0.5h, 0h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 4.5h, 5h, 5.5h, 6h, 6.5h, 7h, 7.5h, 8h, 9h, 10h, 11h, 12h
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nmol/L
Groups:
- Infacort 10 mg: Multi-particulate granules from 1 Infacort 10 mg capsule
- Hydrocortisone: 1 (10 mg) hydrocortisone tablet
Arm/Group | Infacort 10 mg | Hydrocortisone
Number analyzed (Participants) | 14 | 14
hr*nmol/L | 1836.718 (17.8) | 1803.278 (14.6)

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Infacort at Doses of 0.5, 2, 5 and 10 mg
Description: To determine the dose proportionality for Infacort® at doses of 0.5 mg, 2 mg, 5 mg and 10 mg.
Time Frame: -1h, -0.5h, 0h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 4.5h, 5h, 5.5h, 6h, 6.5h, 7h, 7.5h, 8h, 9h, 10h, 11h, 12h
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- Infacort 0.5mg: Multi-particulate granules from 1 (0.5 mg) capsule
  Infacort: Multi-particulate granules
- Infacort 2mg: Multi-particulate granules from 1 (2mg) capsule
  Infacort: Multi-particulate granules
- Infacort 5mg: Multi-particulate granules from 1 (5mg) capsule
  Infacort: Multi-particulate granules
- Infacort 10mg: Multi-particulate granules from 1 (10mg) capsule
  Infacort: Multi-particulate granules
Arm/Group | Infacort 0.5mg | Infacort 2mg | Infacort 5mg | Infacort 10mg
Number analyzed (Participants) | 15 | 15 | 15 | 14
nmol/L | 92.220 (22.9) | 242.798 (16.0) | 424.310 (14.8) | 601.843 (21.5)

5. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Infacort at Doses of 0.5, 2, 5 and 10 mg
Description: To determine the dose proportionality for Infacort® at doses of 0.5 mg, 2 mg, 5 mg and 10 mg.
Time Frame: -1h, -0.5h, 0h, 0.5h, 1h, 1.5h, 2h, 2.5h, 3h, 3.5h, 4h, 4.5h, 5h, 5.5h, 6h, 6.5h, 7h, 7.5h, 8h, 9h, 10h, 11h, 12h
Measure: Median (Standard Deviation); unit: Hours
Arm/Group | Infacort 0.5 mg | Infacort 2 mg | Infacort 5 mg | Infacort 10 mg
Number analyzed (Participants) | 15 | 15 | 15 | 14
Hours | 0.500 (0.2236) | 0.500 (0.3010) | 0.500 (0.3162) | 0.500 (0.4031)

6. Secondary Outcome: Area Under the Curve (AUC0-t) of Infacort at Doses of 0.5, 2, 5 and 10 mg
Description: To determine the dose proportionality for Infacort® at doses of 0.5 mg, 2 mg, 5 mg and 10 mg.
Time Frame: 1 day
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: H*nmol/L
Arm/Group | Infacort 0.5 mg | Infacort 2 mg | Infacort 5 mg | Infacort 10 mg
Number analyzed (Participants) | 14 | 14 | 14 | 14
H*nmol/L | 326.129 (21.3) | 648.407 (16.6) | 1127.579 (15.2) | 1836.718 (17.8)

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) as Assessed by Medical Dictionary for Regulatory Activities (MedDRA) Dictionary, Version 16.0.
Description: To assess the safety and tolerability of Infacort® throughout the study. For a full list of TEAEs per arm, please refer to the Adverse Events section.
Time Frame: 1 day
Measure: Number; unit: TEAEs
Arm/Group | All Study Participants
Number analyzed (Participants) | 16
TEAEs | 7

ADVERSE EVENTS:
Time Frame: From study start (19 July 2013) to completion (9 September 2013)
Arm/Group | Infacort 0.5 mg | Infacort 2 mg | Infacort 5 mg | Infacort 10 mg | Hydrocortisone
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 1/16 | 0/16 | 4/16 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infacort 0.5 mg (N=16) | Infacort 2 mg (N=16) | Infacort 5 mg (N=16) | Infacort 10 mg (N=16) | Hydrocortisone (N=16)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must obtain written consent from the Sponsor prior to any publication of results.